CLINICAL TRIAL: NCT05402397
Title: Losartan and Uric Acid Metabolism in Children With Proteinuric Nephropathies: a Cross-over Randomized Clinical Trail
Brief Title: Losartan and Uric Acid Metabolism in Children With Proteinuric Nephropathies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Principal Investigator, Alejandro Balestracci, Staff Nephrology Unit Hospital General de Niños Pedro de Elizalde, Hospital General de Niños Pedro de Elizalde
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HGNPE 7122
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Uric Acid Nephropathy
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Intervention Model Description: Patients already treated with enalapril will be randomized to receive losartan or enalapril in a cross-over designed study. Those who recruit the inclusion criteria will receive enalapril and/or losartan during a one month period, followed by a 15 days of wash out (under enalapril treatment). On day 46, the second period of 30 days of treatment starts (enalapril or losartan, whichever was not received initially).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enalapril (Active Comparator): Children with proteinuric nephropathies will receive enalapril prior or after a losartan period, according to randomization sequence.
  Enalapril will be given at a dose between 0.1 to 0.4 mg/kg/day (according to the dose that they usually receive), once a day.
  Interventions: Drug: Losartan Potassium
- Losartan (Experimental): Children with proteinuric nephropathies will receive losartan prior or after a enalapril period, according to randomization sequence.
  Losartan will be given at a dose 5 times the dose of enalapril that they usually receive, (with a maximum dose of 1.4 mg/kg/day), once a day.
  Interventions: Drug: Losartan Potassium

INTERVENTIONS:
Drug: Losartan Potassium — Patients will receive losartan potassium for 30 days.

SUMMARY:
The aim of this study is to assess the serum uric-acid lowering effect of losartan in children with proteinuric nephropathies. Patients already treated with enalapril will be randomized to receive losartan and/or enalapril in a cross-over designed study. Those who recruit the inclusion criteria will receive enalapril and/or losartan during a one month period, followed by a 15 days of wash out (under enalapril treatment). On day 46, the second period of 30 days of treatment start (enalapril or losartan, whichever was not received initially). Before randomization, a baseline 24 hours urine and a fasting blood sample will be obtained to assess uric acid excretion and serum uric acid values along with renal function and electrolyte levels. Then, similar determinations will be performed at days 30, 46 and 76.

DETAILED DESCRIPTION:
The working hypothesis is that the administration to losartan reduces significantly the serum uric acid levels in normotensive children with proteinuric nephropathies. The study will consist in a single center cross-over randomized, open label, clinical trial.

Inclusion criteria will be:children with poteinuric nephropathies already treated with enalapril under our care, age between 3 and 12 years and normal blood pressure.

Subjects will be selected by simple probability sampling and after the signature of the assent/informed consent, they will be randomized (blocks of 4 patients, treatment sequence 2:2) to receive a two phases regime of drugs: 1) arm enalapril-losartan, or 2) arm losartan-enalapril. Between phases there will be a 14 days wash out period (during this time patients will continue receiving enalapril, as this drug does not have effect on uric acid metabolism). The dose of enalapril will be that they usually receive, while the dose of losartan will be 5 times the those of enalapril that they usually receive.

Visit Schedule: day 1 (randomization) and 30 for the first drug; 15 days wash out period, day 46 and 76 for the second drug. In each visit a physical examination and blood pressure monitor will be performed, along with the following laboratory parameters: urea, creatinine, electrolytes, uric acid, glycemia, triglycerides, cholesterol and lipopolysaccharides. Simultaneously, in a spot urine morning sample will be determined the levels of uric acid, creatinine, proteinuria y albuminuria.

ELIGIBILITY:
Inclusion Criteria:

* Children with poteinuric nephropathies already treated with enalapril under our care.
* Age between 3 and 12 years.
* Normal blood pressure.

Exclusion Criteria:

* Patients with high blood pressure.
* Post menarche female patients.
* Patients with hypouricemia (< 2 mg/dL).
* Patients treated with diuretics.
* Patients with absolute or relative contraindications to receive RAAS antagonists (glomerular filtration < 30 ml/min/1,73 m2, serum potassium > 5,5 mEq/L).
* Patients with active rheumatic diseases.
* Patients treated with dual blockade of the RAAS (enalapril +losartan).
* Patients treated with calcineurin inhibitors.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Serum uric acid levels after losartan treatment | 30 days
  Patiens will receive a losartan regime after serum uric acid levels will be assessed

SECONDARY OUTCOMES:
Urinary uric acid levels after losartan treatment | 30 days
  Patiens will receive a losartan regime after urinary uric acid levels will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Balestracci, MD, Ph. D., Principal Investigator — Hospital General de Niños Pedro de Elizalde
Locations (1):
- HGNPE, CABA, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Yes
The authors will share the generated data with qualified external researchers during the next 5 years after article publication. All data provided will be anonymized to respect the privacy of patients who have participated in the trail in line with applicable laws and regulations.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: During the next 5 years after article publication.
Access Criteria: Qualified external researchers

REFERENCES:
- [Background] Park JH, Jo YI, Lee JH. Renal effects of uric acid: hyperuricemia and hypouricemia. Korean J Intern Med. 2020 Nov;35(6):1291-1304. doi: 10.3904/kjim.2020.410. Epub 2020 Sep 9. PMID 32872730
- [Background] Wuhl E, Schaefer F. Therapeutic strategies to slow chronic kidney disease progression. Pediatr Nephrol. 2008 May;23(5):705-16. doi: 10.1007/s00467-008-0789-y. Epub 2008 Mar 12. PMID 18335252
- [Background] Weaver DJ Jr. Uric acid and progression of chronic kidney disease. Pediatr Nephrol. 2019 May;34(5):801-809. doi: 10.1007/s00467-018-3979-2. Epub 2018 Jun 21. PMID 29931555
- [Background] Sutton Burke EM, Kelly TC, Shoales LA, Nagel AK. Angiotensin Receptor Blockers Effect on Serum Uric Acid-A Class Effect? J Pharm Pract. 2020 Dec;33(6):874-881. doi: 10.1177/0897190019866315. Epub 2019 Aug 7. PMID 31390929
- [Background] Bryant CE, Rajai A, Webb NJA, Hogg RJ. Effects of losartan and enalapril on serum uric acid and GFR in children with proteinuria. Pediatr Nephrol. 2021 Oct;36(10):3211-3219. doi: 10.1007/s00467-021-05045-4. Epub 2021 Apr 21. PMID 33881639
- [Background] Hamada T, Ichida K, Hosoyamada M, Mizuta E, Yanagihara K, Sonoyama K, Sugihara S, Igawa O, Hosoya T, Ohtahara A, Shigamasa C, Yamamoto Y, Ninomiya H, Hisatome I. Uricosuric action of losartan via the inhibition of urate transporter 1 (URAT 1) in hypertensive patients. Am J Hypertens. 2008 Oct;21(10):1157-62. doi: 10.1038/ajh.2008.245. Epub 2008 Jul 31. PMID 18670416
- [Background] Kubota M. Hyperuricemia in Children and Adolescents: Present Knowledge and Future Directions. J Nutr Metab. 2019 May 2;2019:3480718. doi: 10.1155/2019/3480718. eCollection 2019. PMID 31192008
- [Background] Dang A, Zhang Y, Liu G, Chen G, Song W, Wang B. Effects of losartan and irbesartan on serum uric acid in hypertensive patients with hyperuricaemia in Chinese population. J Hum Hypertens. 2006 Jan;20(1):45-50. doi: 10.1038/sj.jhh.1001941. PMID 16281062
- [Background] Wurzner G, Gerster JC, Chiolero A, Maillard M, Fallab-Stubi CL, Brunner HR, Burnier M. Comparative effects of losartan and irbesartan on serum uric acid in hypertensive patients with hyperuricaemia and gout. J Hypertens. 2001 Oct;19(10):1855-60. doi: 10.1097/00004872-200110000-00021. PMID 11593107